CLINICAL TRIAL: NCT00286741
Title: Can Group Visits Improve Outcomes of Veterans With Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 03-084
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Diabetes; Hypertension
Keywords: Diabetes; Hypertension; Randomized controlled trials; cost-effectiveness; health services
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical group visits (Experimental): Medical group visits
  Interventions: Other: Diabetes Group Management Visits
- Treatment as Usual control (No Intervention): control

INTERVENTIONS:
Other: Diabetes Group Management Visits — Patients meet in groups and receive education about diabetes, reinforcing each other with their own experiences. Each patient also gets medication management by a physician and pharmacist.
  Arms: Medical group visits

SUMMARY:
Background: Diabetes is a common, morbid and expensive disease among veterans. Achieving adequate glycemic control and blood pressure control can reduce the devastating complications of diabetes. Because the majority of patients do not achieve adequate control of blood sugar and blood pressure, innovative strategies to improve control are needed. One strategy with great potential for veterans receiving VA care is the group clinic. Group clinics have been developed over the last 5-10 years, and have been shown to improve clinical outcomes and reduce outpatient utilization in geriatric settings. Group medical clinics involve a cohort of 8-20 patients who have 1-2 hour group visits. These clinics are distinguished from traditional group education visits for diabetes by the fact that these visits involve one physician and one or more additional health care professionals, usually a nurse practitioner and/or a pharmacist, and are designed to make management changes for a number of people with the same disease in a short period of time. The effect of group medical clinics on blood sugar, blood pressure, and the cost of diabetes care, is unknown. Objectives: Our primary objectives in this project are to determine the effectiveness and cost-effectiveness of a group visit intervention in improving rates of control of diabetes and high blood pressure in patients with both illnesses.

DETAILED DESCRIPTION:
Background:

Diabetes is a common, morbid and expensive disease among veterans. Achieving adequate glycemic control and blood pressure control can reduce the devastating complications of diabetes. Because the majority of patients do not achieve adequate control of blood sugar and blood pressure, innovative strategies to improve control are needed. One strategy with great potential for veterans receiving VA care is the group clinic. Group clinics have been developed over the last 5-10 years, and have been shown to improve clinical outcomes and reduce outpatient utilization in geriatric settings. Group medical clinics involve a cohort of 8-20 patients who have 1-2 hour group visits. These clinics are distinguished from traditional group education visits for diabetes by the fact that these visits involve one physician and one or more additional health care professionals, usually a nurse practitioner and/or a pharmacist, and are designed to make management changes for a number of people with the same disease in a short period of time. The effect of group medical clinics on blood sugar, blood pressure, and the cost of diabetes care, is unknown.

Objectives:

Our primary objectives in this project were to determine the effectiveness and cost-effectiveness of a group visit intervention in improving rates of control of diabetes and high blood pressure in patients with both illnesses.

Methods:

We performed a two-site, randomized, controlled trial of group medical visits for diabetes management. Patients were patients in primary care at the Durham or Richmond VAMC's who had inadequate control of both their blood sugar and their blood pressure. We excluded patients with life-limiting illness. Patients randomized to the control arm received usual primary care. Patients randomized to the intervention arm were assigned to attend a group medical clinic every two months for one year. In the clinic, a primary care physician, with the assistance of a nurse and a pharmacist, measured blood pressure at the point of care, reviewed blood sugar logs, and then made all necessary medical changes for patients with diabetes. The primary outcomes were hemoglobin A1c and systolic blood pressure. Additional outcomes will be serum LDL-cholesterol, diabetes-specific quality of life, and health services utilization. Formative evaluation was undertaken to determine the mechanism of the intervention and to prepare for more successful dissemination if the intervention is effective. Formal cost analysis will be performed and cost-effectiveness analysis will be undertaken. All outcomes were measured at baseline, and 6 and 12 months after the beginning of the intervention.

Status:

All patient contact complete. Project is in analysis phase.

ELIGIBILITY:
Inclusion Criteria:

* Primary care at one of two participating sites,
* HbA1c >= 7.5%, Systolic BP > 140 OR Diastolic BP > 90 on 2 consecutive measurements

Exclusion Criteria:

-Primary care provider excludes patient from study, -Patient states that primary care is shared with non-VA primary care provider, -New enrollment in endocrine clinic within the last 6 months, -Patient is reluctant to participate in group visit for any reason, -Reduced life expectancy, as determined by any of the following: -New York Heart Association Class IV congestive heart failure, -Lung disease requiring supplemental oxygen, -End-stage renal disease on dialysis, -Current malignancy with any evidence of disease or currently undergoing chemotherapy or radiation therapy, -Cirrhosis of the liver, or -AIDS (HIV disease does not exclude a patient in the absence of an AIDS diagnosis), -Five or more errors on Short Portable Mental Status Questionnaire, Psychotic illness with hospitalization within three years prior to enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2006-06; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Edelman, MD MHS, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (2):
- United States (2):
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

REFERENCES:
- [Result] Edelman D, Fredrickson SK, Melnyk SD, Coffman CJ, Jeffreys AS, Datta S, Jackson GL, Harris AC, Hamilton NS, Stewart H, Stein J, Weinberger M. Medical clinics versus usual care for patients with both diabetes and hypertension: a randomized trial. Ann Intern Med. 2010 Jun 1;152(11):689-96. doi: 10.7326/0003-4819-152-11-201006010-00001. PMID 20513826
- [Result] Crowley MJ, Melnyk SD, Ostroff JL, Fredrickson SK, Jeffreys AS, Coffman CJ, Edelman D. Can group medical clinics improve lipid management in diabetes? Am J Med. 2014 Feb;127(2):145-51. doi: 10.1016/j.amjmed.2013.09.027. Epub 2013 Oct 15. PMID 24462012
- [Result] Jackson GL, Edelman D, Olsen MK, Smith VA, Maciejewski ML. Benefits of participation in diabetes group visits after trial completion. JAMA Intern Med. 2013 Apr 8;173(7):590-2. doi: 10.1001/jamainternmed.2013.2803. No abstract available. PMID 23478796
- [Result] Crowley MJ, Melnyk SD, Coffman CJ, Jeffreys AS, Edelman D. Impact of baseline insulin regimen on glycemic response to a group medical clinic intervention. Diabetes Care. 2013 Jul;36(7):1954-60. doi: 10.2337/dc12-1905. Epub 2013 Feb 7. PMID 23393214
- [Result] Edelman D, Dolor RJ, Coffman CJ, Pereira KC, Granger BB, Lindquist JH, Neary AM, Harris AJ, Bosworth HB. Nurse-led behavioral management of diabetes and hypertension in community practices: a randomized trial. J Gen Intern Med. 2015 May;30(5):626-33. doi: 10.1007/s11606-014-3154-9. Epub 2015 Jan 8. PMID 25567758

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: control
Period: Overall Study
Arm/Group | Medical Group Visits | Control
Started | 133 | 106
Completed | 122 | 89
Not Completed | 11 | 17

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Medical group visits
  Diabetes Group Management Visits: Patients meet in groups and receive education about diabetes, reinforcing each other with their own experiences. Each patient also gets medication management by a physician and pharmacist.
- Arm 2: control
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 133 | 106 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.4) | 60.8 (10) | 62.0 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 127 | 102 | 229
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 72 | 71 | 143
  White | 57 | 29 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 128 | 103 | 231
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage points
Groups:
- Control: Treatment as Usual Control
Arm/Group | Medical Group Visits | Control
Number analyzed (Participants) | 133 | 106
percentage points | 8.4 (1.3) | 8.7 (1.5)
Statistical Analysis 1: Comparison: Medical Group Visits vs Control; Test type: Superiority or Other; p = 0.15, Mixed Models Analysis

2. Primary Outcome: Systolic Blood Pressure
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Medical Group Visits | Treatment as Usual Control
Number analyzed (Participants) | 133 | 106
mmHg | 140 (14.8) | 147 (13.4)
Statistical Analysis 1: Comparison: Medical Group Visits vs Treatment as Usual Control; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis

3. Secondary Outcome: Cost-effectiveness, Proportion of Patients With LDL < 100, Health Services Utilization, Quality of Life (as Measured by DQoL), Patient Empowerment (as Measured by DES).
Time Frame: one year
Population: Analysis was not performed - project staff and data no longer available.
Arm/Group | Medical Group Visits | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Medical Group Visits | Control
Serious Adverse Events (participants affected / at risk) | 59/133 | 37/106
Other Adverse Events (participants affected / at risk) | 122/133 | 85/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medical Group Visits (N=133) | Control (N=106)
Death (General disorders) | 3 | 1
All-Cause hospitalization (General disorders) | 56 | 36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medical Group Visits (N=133) | Control (N=106)
Hypoglycemia (Endocrine disorders) | 101 | 83 — Patient self-report, or blood glucose measured < 60
Hypotension (Vascular disorders) | 19 | 14 — Systolic Blood Pressure < 100
Lightheadedness (Vascular disorders) | 66 | 62 — Patient self-report
Renal insufficiency (Renal and urinary disorders) | 71 | 51 — Decrease in estimate Glomerular Filtration Rate > 10 ml/min/1.73 m2
Hepatic insufficiency (Hepatobiliary disorders) | 2 | 2 — Aspartate aminotransferase or alanine aminotransferase > 50 U/liter

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes